CLINICAL TRIAL: NCT02020330
Title: An Open-label Randomized Controlled Trial to Evaluate the Effectiveness and Safety of a 3 Day Versus 5 Day Course of Artemether-lumefantrine for the Treatment of Uncomplicated Falciparum Malaria in Myanmar
Brief Title: Optimising Operational Use of Artemether-lumefantrine Comparing 3 Day Versus 5 Day
Acronym: AL3vs5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOCRU1301
Record Dates: First submitted 2013-10-30; First posted 2013-12-24 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Plasmodium Falciparum Infection
Keywords: falciparum, malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL3days (Active Comparator): Artemether-lumefantrine 3 days
  Interventions: Drug: Artemether-lumefantrine 3 days
- AL5days (Experimental): Artemether-lumefantrine 5 days
  Interventions: Drug: Artemether-lumefantrine 5 days

INTERVENTIONS:
Drug: Artemether-lumefantrine 3 days — One tablet contains 20mg artemether and 120mg lumefantrine. The standard regimen is twice daily for 3 days with a delay of at least 8 hours between the first and second dose. It is dosed by weight categories. One gram of fish oil will be given to half of the participants in the 3 days arm.
  Other Names: Coartem®, Novatis, Switzerland
  Arms: AL3days
Drug: Artemether-lumefantrine 5 days — One tablet contains 20mg artemether and 120mg lumefantrine. The experiment regimen is twice daily for 5 days with a delay of at least 8 hours between the first and second dose. It is dosed by weight categories. One gram of fish oil will be given to half of the participants in the 5 days arm.
  Other Names: Coartem®, Novartis, Switzerland
  Arms: AL5days

SUMMARY:
This is a randomised two arm study, comparing artemether-lumefantrine 3 days and 5 days treatment. Patients will be randomised in blocks of ten to one of the two treatment arms. The standard regimen is twice daily for three days with a delay of at least eight hours between the first and second doses. A single of primaquine will be given to all patients on the first day of treatment for gametocytocidal activity. The initial treatment will be given under supervision, all other subsequent doses will be given to the patient to the taken at home. Patients will be followed up for nine visits over forty two days.

DETAILED DESCRIPTION:
* The study will be conducted in 6 village health centres in the Mon and Kayin states
* The patient or parent/guardian (in case of minor or under aged) must personally sign and date the latest approved version of the informed consent form before any study specific procedures are performed
* A case record form will be completed for each patient documenting symptoms prior to clinic attendance, concomitant illness, drug history. Height, weight, vital signs and physical examination findings will be recorded.
* At enrolment (D0) all patients will have the following samples taken:

  * Repeat parasite count (thick and thin films). Treatment should be started without waiting for the result.
  * Filter paper blood blots (3 dots on Whatman 3MM filter paper approx 180-300 µL blood) for parasite genotyping (MSP1, MSP2, GLURP in case of recurrence during follow-up)
  * Haemoglobin
* Laboratory procedures

  * Slide microscopy: Thick and thin blood films stained with Giemsa will be read and counts expressed as the number of parasites per 500 white blood cells
  * Molecular studies: The samples will be used to detect asexual parasites (blood smear, sensitive PCR), parasite population structure (Sequenom genotyping and sequencing), gametocytes (microscopy). The samples will be stored in a cool box and kept maximum 5 days in the field and will be transported to the local laboratory for processing. Plasma and buffy coat will be separated, frozen and stored. The frozen packed red cells will be transported to the molecular laboratory at MORU, Bangkok, Thailand, for sample processing (DNA extraction, quantitative PCRs).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 year
2. Symptomatic malaria infection, i.e. history of fever or presence of fever >37.5°C
3. Microscopic confirmation of asexual stages of P. falciparum (may be mixed with non-falciparum species) with parasitaemia PFT≥5/500 WBC
4. Written informed consent given to participate in the trial

Exclusion Criteria:

1. Pregnancy or lactation (urine test for β HCG to be performed on any woman of child bearing age unless menstruating).
2. Female of 12 to 18 years of age
3. P. falciparum asexual stage parasitaemia greater than or equal to 4% red blood cells (175,000/µL).
4. Signs or symptoms indicative of severe malaria including:

   * Impaired consciousness (Blantyre Coma Score <5 or Glasgow Coma Scale <15)
   * Severe anaemia (Hb% <5 mg/dl)
   * Bleeding disorder -evidenced by epistaxis, bleeding gums, frank haematuria, bleeding from venepuncture sites
   * Respiratory distress
   * Severe jaundice
   * Haemodynamic shock
5. A full course of artemether-lumefantrine treatment in the previous 28 days
6. Known hypersensitivity to artemisinins - defined as history of erythroderma/other severe cutaneous reaction, angioedema or anaphylaxis
7. History of splenectomy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-03-25 (Actual)

PRIMARY OUTCOMES:
proportion of patients with detectable parasitaemia | On day 5 and day 7
  Assessed by sensitive PCR on days 5 and 7 after treatment

SECONDARY OUTCOMES:
Parasitaemia clearance time | On day 3 and Day 5
  Assessed by sensitive PCR on D3 in the 3 day arm and D5 in the 5 day arm
Gametocyte carriage rates | Day 7
artemether-lumefantrine tolerability | 5 days
  Tolerability of artemether-lumefantrine will be assessed by comparing the proportion of patients with anorexia, nausea, vomiting, abdominal pain and other symptoms of administration between the intervention arm and the control arm
Comparison of effectiveness | Day 42
  Comparison of effectiveness uncorrected and corrected will be assessed by PCR genotyping
concentrations of lumefantrine | Day 7
Haematological recovery rate | Day 28
  Assessed by comparing hemoglobin between baseline and after treatment at day 28
Incidence of vivax malaria relapses | 42 days
  Assessed by the microscopist find malaria smear positive within the follow up period
Comparison of addition of food supplement (fish oil) | day 3 to day 21
  Assessed by comparing lumefantrine concentration on day 7 and proportion of patients with detectable parasitaemia by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Frank Smithuis, MD, Principal Investigator — Myanmar Oxford Clinical Research Unit
Locations (1):
- Medical Action Myanmar, Yangon, Burma

REFERENCES:
- [Derived] Tun KM, Jeeyapant A, Myint AH, Kyaw ZT, Dhorda M, Mukaka M, Cheah PY, Imwong M, Hlaing T, Kyaw TH, Ashley EA, Dondorp A, White NJ, Day NPJ, Smithuis F. Effectiveness and safety of 3 and 5 day courses of artemether-lumefantrine for the treatment of uncomplicated falciparum malaria in an area of emerging artemisinin resistance in Myanmar. Malar J. 2018 Jul 11;17(1):258. doi: 10.1186/s12936-018-2404-4. PMID 29996844